CLINICAL TRIAL: NCT01820065
Title: A Long-term Evaluation of Single-piece Hydrophobic Acrylic Intraocular Lens Implantation on the Development of Posterior Capsule Opacification
Brief Title: Long-term Evaluation of Single-piece ACrysof IOL Implantation on Development of Posterior Capsule Opacification
Status: Completed | Type: Observational
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Principal Investigator, Abhay R. Vasavada, Director, Iladevi Cataract and IOL Research Center, Iladevi Cataract and IOL Research Center
Other Study IDs: 05-003
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Posterior Capsule Opacification After Phacoemulsification and IOL Implantation
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients undergoing phacoemulsification: Patients undergoing phacoemulsification for age-related cataract with implantation of a single-piece Acrysof IOL (SN60AT)
  Interventions: Procedure: Cataract surgery with IOL implantation

INTERVENTIONS:
Procedure: Cataract surgery with IOL implantation — Phacoemulsification with implantation of single piece Acrysof IOL

SUMMARY:
Although contemporary cataract surgery has made tremendous strides in technological advancement, posterior capsular opacification (PCO) is still the most frequent long-term complication leading to decreased visual functions and thereby dissatisfying results. A great deal of effort has been made to develop new ways to prevent the formation of PCO. A key factor, widely discussed in literature, is the material and design of the intraocular lense (IOL) edge that can lead to PCO prevention. It is still not clear whether the sharp-edged IOL produces less PCO because of its optic geometry alone or whether the biomaterial contributes to the inhibition of PCO. With the clinical introduction of the single-piece acrylic hydrophobic IOLs with some optic and haptic design differences compared with three-piece acrylic hydrophobic IOLs, it has become possible to determine the influence of IOL material and design on PCO prevention. It is well established that the development of PCO is a dynamic process and that a longer follow-up time is correlated with a higher degree of PCO. So far, there have been prospective clinical studies on the clinical results of single and three-piece acrylic hydrophobic foldable IOLs. However, the question as to as to whether the PCO further increases or becomes stable or regresses on a long-term basis has not yet been answered. Since there is paucity of available literature that prospectively evaluates the development of PCO with the implantation of the single-piece SN60AT hydrophobic acrylic IOL on a long-term basis, the investigators decided to observe the degree of development of PCO at 5 years after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with uncomplicated age-related cataract who were otherwise healthy

Exclusion Criteria:

* a history of diabetes mellitus (DM),
* patients with glaucoma,
* high myopia (axial length > 27.0 mm),
* pseudoexfoliation,
* traumatic cataract,
* subluxated cataract,
* previous ocular surgeries, and
* allergy to dilating drops.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing phacoemulsification for age-related uncomplicated phacoemulsification
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2005-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Posterior Capsule Opacification | 5 years followup
  Evaluation of PCO (EPCO) scores in the area of the intraocular lens (IOL) optic and in the central 3mm zone at 5 years after surgery

SECONDARY OUTCOMES:
EPCO Score and EPCO area with total on and part on anterior capsulorhexis cover over optic | 5 years postoperatively

OTHER OUTCOMES:
Change in PCO at different followup intervals | upto 5 years postoperatively
  Change in PCO observed from 1 month to 1 year, 1 year to 3 years, and 3 years to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Abhay R Vasavada, MS, FRCS, Principal Investigator — Iladevi Cataract & IOL Research Centre; Abhay R Vasavada, MS,FRCS, Principal Investigator — Iladevi Cataract & IOL Research Centre
Locations (1):
- Iladevi Cataract & IOL Research Centre, Ahmedabad, Gujarat, India